CLINICAL TRIAL: NCT02467842
Title: A Multi-center, Randomized, Double-blind Phase III Clinical Trial to Assess the Immunogenicity and Safety of Quadrivalent Inactivated Cell Culture-derived Influenza Vaccine in Adults and Elderly Subjects
Brief Title: Immunogenicity and Safety of Quadrivalent Influenza Vaccine (NBP607-QIV) in Adults and Elderly Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SK Chemicals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NBP607-QIV_FluA_III_2014
Record Dates: First submitted 2015-06-03; First posted 2015-06-10 (Estimated); Results first posted 2020-05-08 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2015-06

CONDITIONS: Influenza
Keywords: Influenza vaccine; Quadrivalent; Inactivated cell culture-derived
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NBP607-QIV (Experimental): Participants aged 19 years and older received a 0.5mL single intramuscular dose of Quadrivalent Inactivated Cell Culture-derived Influenza Vaccine containing 4 virus strains; A/H1N1, A/H3N2, B/Yamagata, B/Victoria on Day 0
  Interventions: Biological: NBP607-QIV
- NBP607-Y (Active Comparator): Participants aged 19 years and older received a 0.5mL single intramuscular dose of Trivalent Inactivated Cell Culture-derived Influenza Vaccine containing 3 virus strains; A/H1N1, A/H3N2, B/Yamagata on Day 0
  Interventions: Biological: NBP607-Y
- NBP607-V (Active Comparator): Participants aged 19 years and older received a 0.5mL single intramuscular dose of Trivalent Inactivated Cell Culture-derived Influenza Vaccine containing 3 virus strains; A/H1N1, A/H3N2, B/Victoria on Day 0
  Interventions: Biological: NBP607-V

INTERVENTIONS:
Biological: NBP607-QIV — Quadrivalent Inactivated Cell Culture-derived Influenza Vaccine containing 4 virus strains; A/H1N1, A/H3N2, B/Yamagata, B/Victoria
  Arms: NBP607-QIV
Biological: NBP607-Y — Trivalent Inactivated Cell Culture-derived Influenza Vaccine containing 3 virus strains; A/H1N1, A/H3N2, B/Yamagata
  Arms: NBP607-Y
Biological: NBP607-V — Trivalent Inactivated Cell Culture-derived Influenza Vaccine containing 3 virus strains; A/H1N1, A/H3N2, B/Victoria
  Arms: NBP607-V

SUMMARY:
All participants received a single dose of their assigned vaccine on Day 0. They were followed up for immunogenicity and safety through Day 21 post-vaccination. Serious adverse events were collected for 6 months post-vaccination.

DETAILED DESCRIPTION:
In a randomized controlled phase III trial undertaken in 10 university hospitals of South Korea, adults and elderly subjects were randomly assigned in a 2:1:1 ratio to NBP607-QIV versus cell culture-based trivalent inactivated influenza vaccine (TIV), NBP607-Y and NBP607-V. Immunogenicity was assessed 3 weeks after vaccination by hemagglutination inhibition (HI) assay. Safety was assessed for 6 months post-vaccination: solicited adverse events for 7 days, unsolicited adverse events (AEs) for 21 days and serious adverse events (SAE) for 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 19 years and older
* Those who are able to comply with the requirements for the study
* If women, a negative pregnancy test and willingness to use birth control measures for the entire study duration

Exclusion Criteria:

* Disorders in immune function
* Any malignancy or lymphoproliferative disorder
* History of Guillain-Barré syndrome
* Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time
* Experience of fever (>38.0 ℃) within 24 hours following vaccination
* Body temperature >38.0 ℃ at the vaccination day
* Concomitant medications/therapy such as immunosuppressants or immune modifying drugs, systemic corticosteroids, immunoglobulins, blood or blood- derived products within 3 months
* Influenza vaccination within 6 months
* Subjects who have participated in other interventional study within 4 weeks
* Any vaccination within 1 month
* Those who are planning to receive any vaccine within 1 month from the study vaccine
* Individuals with any serious chronic or progressive disease
* Pregnant or breast-feeding women
* Any other reason that in the opinion of the investigator might interfere with the study

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1503 (Actual)
Dates: Start 2014-10; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Woo Joo Kim, MD, PhD, Study Chair — Korea University Guro Hospital; Won Suk Choi, MD, PhD, Principal Investigator — Korea University; Seong-Heon Wie, MD, PhD, Principal Investigator — Catholic University St. Vincent's Hospital; Jin Soo Lee, MD, PhD, Principal Investigator — Inha University Hospital; Jacob Lee, MD, PhD, Principal Investigator — Hallym University Kangnam Sacred Heart Hospital; Shin Woo Kim, MD, PhD, Principal Investigator — Kyungpook University Hospital; Hye Won Jeong, MD, Principal Investigator — Chungbuk University Hospital; Sook-In Jung, MD, Principal Investigator — Chonnam University Hospital; Yeon-Sook Kim, MD, PhD, Principal Investigator — Chungnam University Hospital; Heung Jeong Woo, MD, PhD, Principal Investigator — Hallym University Dongtan Sacred Heart Hospital

REFERENCES:
- [Result] Choi WS, Noh JY, Song JY, Cheong HJ, Wie SH, Lee JS, Lee J, Kim SW, Jeong HW, Jung SI, Kim YS, Woo HJ, Kim KH, Kim H, Kim WJ. Immunogenicity and safety of a cell culture-derived inactivated quadrivalent influenza vaccine (NBP607-QIV): A randomized, double-blind, multi-center, phase III clinical trial in adults and elderly subjects. Hum Vaccin Immunother. 2017 Jul 3;13(7):1653-1660. doi: 10.1080/21645515.2017.1297351. Epub 2017 Apr 13. PMID 28406746

RESULTS

PARTICIPANT FLOW:
Groups:
- NBP607-QIV: Participants received a 0.5mL single intramuscular dose on Day 0
  NBP607-QIV: Quadrivalent Inactivated Cell Culture-derived Influenza Vaccine containing 4 virus strains; A/H1N1, A/H3N2, B/Yamagata, B/Victoria
- NBP607-Y: Participants received a 0.5mL single intramuscular dose on Day 0
  NBP607-Y: Trivalent Inactivated Cell Culture-derived Influenza Vaccine containing 3 virus strains; A/H1N1, A/H3N2, B/Yamagata
- NBP607-V: Participants received a 0.5mL single intramuscular dose on Day 0
  NBP607-V: Trivalent Inactivated Cell Culture-derived Influenza Vaccine containing 3 virus strains; A/H1N1, A/H3N2, B/Victoria
Period: Overall Study
Arm/Group | NBP607-QIV | NBP607-Y | NBP607-V
Started | 752 | 373 | 378
Completed | 752 | 373 | 378
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- NBP607-QIV: Participants aged 19 years and older received a 0.5mL single intramuscular dose on Day 0
  NBP607-QIV: Quadrivalent Inactivated Cell Culture-derived Influenza Vaccine containing 4 virus strains; A/H1N1, A/H3N2, B/Yamagata, B/Victoria
- NBP607-Y: Participants aged 19 years and older received a 0.5mL single intramuscular dose on Day 0
  NBP607-Y: Trivalent Inactivated Cell Culture-derived Influenza Vaccine containing 3 virus strains; A/H1N1, A/H3N2, B/Yamagata
- NBP607-V: Participants aged 19 years and older received a 0.5mL single intramuscular dose on Day 0
  NBP607-V: Trivalent Inactivated Cell Culture-derived Influenza Vaccine containing 3 virus strains; A/H1N1, A/H3N2, B/Victoria
- Total: Total of all reporting groups
Arm/Group | NBP607-QIV | NBP607-Y | NBP607-V | Total
Number analyzed (Participants) | 752 | 373 | 378 | 1503
Age, Customized [Count of Participants; unit: Participants]
  19 to 59 years old | 599 | 299 | 305 | 1203
  60 years old and older | 153 | 74 | 73 | 300
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 476 | 238 | 233 | 947
  Male | 276 | 135 | 145 | 556

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean HI Titers (GMTs) After Vaccination in All Subjects
Description: GMTs of anti-influenza antibodies were measured for 4 strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. For each A strain, the titers were made with the pooled TIV group (NBP60-Y and NBP607-V).
  For each A strain, the comparion was made with the pooled TIV groups (Y+V/QIV). For each B strain, the comparison was made with the corresponding TIV group(i.e. for B/Yamagata, Geometric Mean Titer Ratio (GMR) is Y/QIV).
Time Frame: At Day 21 post vaccination.
Population: Per Protocol Set.
Measure: Geometric Mean (95% Confidence Interval); unit: titers
Arm/Group | NBP607-QIV | NBP607-Y | NBP607-V
Number analyzed (Participants) | 748 | 371 | 376
titers
  A/H1N1 | 329.76 [309.17 to 351.71] | 334.98 [313.91 to 357.47] | 334.98 [313.91 to 357.47]
  A/H3N2 | 401.21 [378.87 to 424.87] | 377.34 [356.47 to 399.44] | 377.34 [356.47 to 399.44]
  B/Yamagata | 163.74 [156.11 to 171.73] | 144.65 [135.54 to 154.37] | 123.08 [115.39 to 131.28]
  B/Victoria | 124.82 [119.16 to 130.75] | 93.29 [87.43 to 99.53] | 112.20 [105.20 to 119.66]
Statistical Analysis 1: Comparison: NBP607-QIV vs NBP607-Y vs NBP607-V; GMR of A/H1N1 strain (GMTs of pooled TIV/QIV); Test type: Non-Inferiority — Non-inferiority of GMTs was concluded if the upper limit of 95% confidence interval of the GMR (active comparator/experimental) was ≤1.5 for each strain; GMR (pooled TIV/QIV) = 1.02, 95% CI 2-sided [0.94 to 1.10]
Statistical Analysis 2: Comparison: NBP607-QIV vs NBP607-Y vs NBP607-V; GMR of A/H3N2 strain (GMTs of pooled TIV/QIV); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMR (pooled TIV/QIV) = 0.94, 95% CI 2-sided [0.87 to 1.01]
Statistical Analysis 3: Comparison: NBP607-QIV vs NBP607-Y; GMR of B/Yamagata strain (GMTs of TIV/QIV); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMR (TIV/QIV) = 0.88, 95% CI 2-sided [0.82 to 0.95]
Statistical Analysis 4: Comparison: NBP607-QIV vs NBP607-V; GMR of A/H1N1 strain (GMTs of TIV/QIV); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; GMR (TIV/QIV) = 0.90, 95% CI 2-sided [0.83 to 0.97]

2. Primary Outcome: Seroconversion Rate (SCR) After Vaccination in All Subjects
Description: SCR was measured for 4 strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. Seroconversion was defined as the proportion of subjects who met either (1) post-vaccination HI titer of ≥ 1:40 for subjects with pre-vaccination HI titer of <1:10 or (2) Four-fold increase in post-vaccination HI titer for subjects with pre-vaccination HI titer of ≥ 1:10
  For each A strain, the comparion was made with the pooled TIV groups (Y+V minus QIV). For each B strain, the comparison was made with the corresponding TIV group(i.e. for B/Yamagata, Difference of SCR (Diff.SCR) is Y minus QIV).
Time Frame: At Day 21 post vaccination.
Population: Per protocol set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NBP607-QIV | NBP607-Y | NBP607-V
Number analyzed (Participants) | 748 | 371 | 376
percentage of participants
  A/H1N1 | 52.41 [48.83 to 55.99] | 52.56 [47.48 to 57.64] | 50.27 [45.21 to 55.32]
  A/H3N2 | 51.20 [47.62 to 54.79] | 46.09 [41.02 to 51.16] | 46.28 [41.24 to 51.32]
  B/Yamagata | 43.72 [40.16 to 47.27] | 36.66 [31.75 to 41.56] | 24.73 [20.37 to 29.10]
  B/Victoria | 55.75 [52.19 to 59.31] | 43.13 [38.09 to 48.17] | 52.66 [47.61 to 57.71]
Statistical Analysis 1: Comparison: NBP607-QIV vs NBP607-Y vs NBP607-V; Diff. SCR of A/H1N1 strain (SCR of pooled TIV minus QIV); Test type: Non-Inferiority — Non-inferiority of SCR was concluded if the upper limit of 95% confidence interval for Diff. SCR (active comparator minus experimental) ≤10% for each strain; Difference in percentage = -1.00, 95% CI 2-sided [-6.07 to 4.06]
Statistical Analysis 2: Comparison: NBP607-QIV vs NBP607-Y vs NBP607-V; Diff. SCR of A/H3N2 strain (SCR of pooled TIV minus QIV); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in percentage = -5.02, 95% CI 2-sided [-10.08 to 0.04]
Statistical Analysis 3: Comparison: NBP607-QIV vs NBP607-Y; Diff. SCR of B/Yamaga strain (SCR of TIV minus QIV); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in percentage = -7.06, 95% CI 2-sided [-13.12 to -1.00]
Statistical Analysis 4: Comparison: NBP607-QIV vs NBP607-V; Diff. SCR of B/Victoria (SCR of TIV minus QIV); Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Difference in percentage = -3.09, 95% CI 2-sided [-9.26 to 3.09]

3. Primary Outcome: Seroprotection Rate (SPR) of NBP607-QIV in the Elderly Subject Aged ≥60 Years
Description: SPR of NBP607-QIV was measured for 4 strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. Seroprotection was defined as the proportion of subjects whose post-vaccination HI titer increased to ≥1:40.
Time Frame: At Day 21 post vaccination.
Population: Per protocol set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- NBP607-QIV: Participants aged 60 years and older received a 0.5mL single intramuscular dose on Day 0
  NBP607-QIV: Quadrivalent Inactivated Cell Culture-derived Influenza Vaccine containing 4 virus strains; A/H1N1, A/H3N2, B/Yamagata, B/Victoria
Arm/Group | NBP607-QIV
Number analyzed (Participants) | 152
percentage of participants
  A/H1N1 | 92.76 [88.64 to 96.88]
  A/H3N2 | 98.68 [96.87 to 100.00]
  B/Yamagata | 94.08 [90.33 to 97.83]
  B/Victoria | 96.05 [92.96 to 99.15]

4. Primary Outcome: Seroconversion Rate (SCR) of NBP607-QIV in the Elderly Subject Aged ≥60 Years
Description: SCR was measured for 4 strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. Seroconversion was defined as the proportion of subjects who met either (1) post-vaccination HI titer of ≥ 1:40 for subjects with pre-vaccination HI titer of <1:10 or (2) Four-fold increase in post-vaccination HI titer for subjects with pre-vaccination HI titer of ≥ 1:10
Time Frame: At Day 21 post vaccination.
Population: Per protocol set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NBP607-QIV
Number analyzed (Participants) | 152
percentage of participants
  A/H1N1 | 52.63 [44.69 to 60.57]
  A/H3N2 | 42.11 [34.26 to 49.95]
  B/Yamagata | 43.42 [35.54 to 51.30]
  B/Victoria | 59.87 [52.08 to 67.66]

5. Primary Outcome: Geometric Mean Ratio (GMR) of NBP607-QIV in the Elderly Subject Aged ≥60 Years
Description: GMR was measured for 4 strains: A/H1N1, A/H3N2, B/Victoria, and B/Yamagata. GMR was defined as the fold-rise of the geometric mean HI titer from pre- to post-vaccination.
Time Frame: At Day 21 post vaccination.
Population: Per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | NBP607-QIV
Number analyzed (Participants) | 152
ratio
  A/H1N1 | 4.07 [3.39 to 4.90]
  A/H3N2 | 3.27 [2.69 to 3.97]
  B/Yamagata | 2.99 [2.59 to 3.44]
  B/Victoria | 4.61 [3.91 to 5.42]

6. Secondary Outcome: Geometric Mean HI Titers (GMTs) of Each B Strain After Vaccination in All Subjects
Description: GMTs of anti-influenza antibodies were measured for B strains: B/Victoria, and B/Yamagata.
  For each B strain, the comparison was made with the TIV group which did not contain the correponding B strain (i.e. for B/Yamagata, Geometric Mean Titer Ratio (GMR) is V/QIV).
Time Frame: At Day 21 post vaccination.
Population: Per protocol set.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | NBP607-QIV | NBP607-Y | NBP607-V
Number analyzed (Participants) | 748 | 371 | 376
titer
  B/Yamagata | 163.74 [156.11 to 171.73] | 144.65 [135.54 to 154.37] | 123.08 [115.39 to 131.28]
  B/Victoria | 124.82 [119.16 to 130.75] | 93.29 [87.43 to 99.53] | 112.20 [105.20 to 119.66]
Statistical Analysis 1: Comparison: NBP607-QIV vs NBP607-V; GMR of B/Yamagata strain (GMTs of TIV/QIV); Test type: Superiority — Superiority of GMTs was concluded if the upper limit of 95% confidence interval for GMR (active comparator/experimental) was ≤1.0 for each B strain; GMR (TIV/QIV) = 0.75, 95% CI 2-sided [0.70 to 0.81]
Statistical Analysis 2: Comparison: NBP607-QIV vs NBP607-Y; GMR of B/Victoria (GMTs of TIV/QIV); Test type: Superiority — [test comment as in outcome 6, analysis 1]; GMR (TIV/QIV) = 0.75, 95% CI 2-sided [0.69 to 0.81]

7. Secondary Outcome: Seroconversion Rate (SCR) of B Strain After Vaccination in All Subjects
Description: SCR was measured for each B strain: B/Victoria, and B/Yamagata. Seroconversion was defined as the proportion of subjects who met either (1) post-vaccination HI titer of ≥ 1:40 for subjects with pre-vaccination HI titer of <1:10 or (2) Four-fold increase in post-vaccination HI titer for subjects with pre-vaccination HI titer of ≥ 1:10
Time Frame: At Day 21 post vaccination.
Population: Per protocol set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NBP607-QIV | NBP607-Y | NBP607-V
Number analyzed (Participants) | 748 | 371 | 376
percentage of participants
  B/Yamagata | 43.72 [40.16 to 47.27] | 36.66 [31.75 to 41.56] | 24.73 [20.37 to 29.10]
  B/Victoria | 55.75 [52.19 to 59.31] | 43.13 [38.09 to 48.17] | 52.66 [47.61 to 57.71]
Statistical Analysis 1: Comparison: NBP607-QIV vs NBP607-V; Diff. SCR of B/Yamaga strain (SCR of TIV minus QIV); Test type: Superiority — Superiority was concluded if the upper limit of 95% confidence interval for Diff. SCR (active comparator-experimental) was ≤0% in each B strain; Difference in percentage = -18.98, 95% CI 2-sided [-24.61 to -13.36]
Statistical Analysis 2: Comparison: NBP607-QIV vs NBP607-Y; Diff. SCR of B/Victoria strain (SCR of TIV minus QIV); Test type: Superiority — [test comment as in outcome 7, analysis 1]; Difference in percentage = -12.62, 95% CI 2-sided [-18.79 to -6.45]

8. Secondary Outcome: Seroprotection Rate (SPR) of NBP607-QIV in the Adults Aged 19 to 59 Years
Description: as for outcome 3
Time Frame: At Day 21 post vaccination.
Population: Per protocol set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- NBP607-QIV: Participants aged 19 to 59 years received a 0.5mL single intramuscular dose on Day 0
  NBP607-QIV: Quadrivalent Inactivated Cell Culture-derived Influenza Vaccine containing 4 virus strains; A/H1N1, A/H3N2, B/Yamagata, B/Victoria
Arm/Group | NBP607-QIV
Number analyzed (Participants) | 596
percentage of participants
  A/H1N1 | 98.32 [97.29 to 99.35]
  A/H3N2 | 99.50 [98.93 to 100.00]
  B/Yamagata | 98.49 [97.51 to 99.47]
  B/Victoria | 99.16 [98.43 to 99.89]

9. Secondary Outcome: Seroconversion Rate (SCR) of NBP607-QIV in the Adults Aged 19 to 59 Years
Description: as for outcome 4
Time Frame: At Day 21 post vaccination.
Population: Per protocol set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | NBP607-QIV
Number analyzed (Participants) | 596
percentage of participants
  A/H1N1 | 52.35 [48.34 to 56.36]
  A/H3N2 | 53.52 [49.52 to 57.53]
  B/Yamagata | 43.79 [39.81 to 47.78]
  B/Victoria | 54.70 [50.70 to 58.69]

10. Secondary Outcome: Geometric Mean Ratio (GMR) of NBP607-QIV in the Subjects Aged 19 to 59 Years
Description: as for outcome 5
Time Frame: At Day 21 post vaccination.
Population: Per protocol set
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | NBP607-QIV
Number analyzed (Participants) | 596
ratio
  A/H1N1 | 4.83 [4.29 to 5.43]
  A/H3N2 | 3.80 [3.45 to 4.18]
  B/Yamagata | 3.21 [2.95 to 3.50]
  B/Victoria | 4.08 [3.73 to 4.46]

ADVERSE EVENTS:
Time Frame: 1) Incidence rate of solicited adverse events (AEs) occured within 7 days after test drug or comparator vaccination 2) Incidence rate of unsolicited AEs occured within 21 days after test drug or comparator vaccination 3) Incidence rate of serious adverse events (SAEs) occured within 6 months after test drug or comparator vaccination
Arm/Group | NBP607-QIV | NBP607-Y | NBP607-V
All-Cause Mortality (participants affected / at risk) | 0/752 | 0/373 | 0/378
Serious Adverse Events (participants affected / at risk) | 9/752 | 3/373 | 3/378
Other Adverse Events (participants affected / at risk) | 364/752 | 154/373 | 151/378
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NBP607-QIV (N=752) | NBP607-Y (N=373) | NBP607-V (N=378)
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Mild Severity, recovered, unrelated to NBP607-QIV
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
acute abdomen (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
colon operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
prostatic specific antigen increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NBP607-QIV (N=752) | NBP607-Y (N=373) | NBP607-V (N=378)
Tenderness (General disorders) | 207 (207) | 84 (84) | 81 (81)
Pain (General disorders) | 198 (198) | 70 (70) | 71 (71)
Redness/erythema (Skin and subcutaneous tissue disorders) | 44 (44) | 18 (18) | 14 (14)
Induration/swelling (General disorders) | 14 (14) | 8 (8) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 130 (130) | 58 (58) | 55 (55)
Fatigue/Malaise (General disorders) | 101 (101) | 71 (71) | 60 (60)
Headache (Nervous system disorders) | 71 (71) | 35 (35) | 38 (38)
Diarrhea (Gastrointestinal disorders) | 25 (25) | 9 (9) | 12 (12)
Vomiting (Gastrointestinal disorders) | 9 (9) | 1 (1) | 2 (2)
Fever (General disorders) | 3 (3) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes